CLINICAL TRIAL: NCT03821129
Title: GORE® CARDIOFORM Septal Occluder and Antiplatelet Medical Management for Reduction of Recurrent Stroke in Patients With Patent Foramen Ovale (PFO): the REDUCE Post Approval Study
Acronym: REDUCE PAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GSO 18-01
Record Dates: First submitted 2019-01-15; First posted 2019-01-29 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Stroke; PFO - Patent Foramen Ovale
Keywords: Occluder; Patent Foramen Ovale; PFO; Stroke; Gore Septal Occluder
MeSH Terms: conditions — Stroke; Foramen Ovale, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- GORE® CARDIOFORM Septal Occluder (Other): Single Arm Commercially available GORE® CARDIOFORM Septal Occluder
  Interventions: Device: PFO closure with GORE® CARDIOFORM Septal Occluder

INTERVENTIONS:
Device: PFO closure with GORE® CARDIOFORM Septal Occluder — PFO closure with GORE® CARDIOFORM Septal Occluder in patients with ischemic stroke

SUMMARY:
This study will assess the safety and effectiveness of GORE® CARDIOFORM Septal Occluder in a post approval setting and evaluate the quality of operator education and training and transferability of trial experience to a post-market setting.

DETAILED DESCRIPTION:
A maximum of 636 adult subjects will be enrolled at up to 40 U.S. centers. Subjects will have follow-up at 1 month, 6 months, 12 months and annually thereafter through 5 years post implant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with an ischemic stroke presumed to be an embolic stroke of undetermined source (ESUS) verified by a neurologist within the last 365 days prior to enrollment.
* Presence of Patent Foramen Ovale (PFO), as determined initially by positive bubble study utilizing transesophageal echocardiography (TEE) and/or transcranial Doppler (TCD), demonstrating spontaneous right-to-left shunting or right-to-left shunting during Valsalva maneuver.
* Patient is able to tolerate antiplatelet therapy
* Note: Additional Inclusion Criteria may apply

Exclusion Criteria:

* History of or ongoing atrial fibrillation/flutter
* Other co-morbidities including, but not limited to, mural thrombus, dilated cardiomyopathy, cardiac prosthetics (valves), severe native valve disease (including mitral valve stenosis), severe ventricular wall motion abnormalities, aortic dissection, significant atherosclerosis, vasculitis, pre-existing non-vascular neurologic disorders, pulmonary arteriovenous malformations, prior intracranial hemorrhage, severe disability related to prior stroke, autoimmune disorders that would increase the risk of stroke or thromboembolism, or associated with increased risk of infection or procedural complications, in the opinion of the investigator, left ventricular ejection fraction of <40%, coexistent cause or intra-cardiac shunting (e.g. VSD or ASD)
* Previous Myocardial Infarction
* Rankin Scale sore greater than or equal to 3 at the time of procedure
* Active infection that cannot be treated successfully prior to enrollment
* Neurological deficits not due to stroke that may affect the patient's neurologic assessments
* Evidence of hypercoagulable state, Uncontrolled diabetes mellitus, uncontrolled systemic hypertension or pulmonary hypertension at the time of screening or procedure
* Sensitivity or contraindication to all proposed medical treatments or any device components
* Pregnant, lactating, or intent on becoming pregnant through 24 months after enrollment.
* Indications outside the parameters accepted for placement of GSO, including extensive congenital cardiac anomalies and defect diameters considered too large for closure with the device.
* Atrial septal anatomy that is expected to necessitate placement of more than one GORE® CARDIOFORM Septal Occluder
* Need for concomitant procedure(s) that may confound detection of adverse events related to device placement
* Note: Additional Exclusion Criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Estimated)
Dates: Start 2019-07-25 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with recurrent ischemic stroke post study device implant (Primary Effectiveness Outcome) | 24 months
  Proportion of subjects with recurrent ischemic stroke post study device implant
Proportion of subjects with device- or procedure-related serious adverse events at 30 days (Primary Safety Endpoint) | 30 days
  Device- or procedure- related serious adverse events post study device implant

SECONDARY OUTCOMES:
Effective PFO Closure defined as complete PFO closure or a trivial or small residual shunt by Echocardiographic assessment | 12 months
  Complete PFO closure or a trivial or small residual shunt
  Proportion of subjects with complete PFO closure or a trivial or small residual shunt
Clinically Significant New Atrial Arrhythmia | 60 months
  Any new atrial fibrillation or flutter
Clinically Significant New Atrial Arrhythmia by Age | 60 months
  Any new atrial fibrillation or flutter in patients greater and less than 60 years of age
Residual Shunt Characterization via assessment of shunt in patients by Echo | 24 months
  Assessment of shunt in patients by Echo
Technical Success defined as successful delivery and retention of the GSO device based on physician reporting | Index procedure
  Successful delivery and retention of the GSO device
Procedural Success defined as successful implantation of the GSO device with no reported in-hospital Serious Adverse Events (SAEs) | Enrollment through discharge, approximately 1 day
  Successful implantation of the GSO device with no reported in-hospital SAEs

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - St. Mary's Hospital, Tucson, Arizona
  - Scripps Health La Jolla, La Jolla, California
  - Loma Linda University Health, Loma Linda, California
  - University of California - San Francisco, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - South Denver Cardiology Associates, Littleton, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Baptist Health Jacksonville, Jacksonville, Florida
  - Naples Community Hospital, Naples, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Northwestern University, Evanston, Illinois
  - University of Iowa Hospitals & Clinic, Iowa City, Iowa
  - Catholic Health Initiatives- Iowa Corp dba Iowa Heart, West Des Moines, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Covenant Medical Center, Inc., Saginaw, Michigan
  - University of Minnesota, Edina, Minnesota
  - Minneapolis Heart Institute Foundation - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Jersey Shore University / Hackensack UMC, Freehold, New Jersey
  - Research Foundation SUNY Buffalo, Buffalo, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - Atrium Health, Charlotte, North Carolina
  - Providence Heart & Vascular Institute, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Tennova Healthcare, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine-Houston, Houston, Texas
  - The Methodist Hospital - Houston, Houston, Texas
  - Methodist Healthcare Systems of San Antonio d/b/a Methodist Hospital, San Antonio, Texas
  - Baylor Scott & White Memorial Hospital, Temple, Texas
  - St. Marks Hospital, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Multicare Health Tacoma-Multicare Institute for Research & Innovation, Tacoma, Washington
  - Charleston Area Medical Center (CAMC), Charleston, West Virginia
  - Aurora Health Care, Metro Inc., Milwaukee, Wisconsin
  - Medical College of Wisconsin, Inc., Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No